CLINICAL TRIAL: NCT05305196
Title: The Effects of Eccentric-focused Exercise on Shoulder Mobility, Rotator Cuff Strength, Pain and Dysfunction, Scapular Kinematics and Muscle Activation in Symptomatic Overhead Athletes With Posterior Shoulder Tightness
Brief Title: The Effects of Eccentric-focused Exercise on Posterior Shoulder Tightness in Symptomatic Overhead Athletes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YM110191F
Record Dates: First submitted 2022-02-17; First posted 2022-03-31 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-03

CONDITIONS: Posterior Shoulder Tightness
Keywords: Posterior shoulder tightness; Eccentric exercise; Shoulder impingement syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Muscle Stretching Exercises; Massage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eccentric-focused exercise group (Experimental): Three eccentric-focused exercises addition to the general treatment group
  Interventions: Other: Eccentric-focused exercises; Other: Stretching exercises; Other: Hot pack; Other: Massage
- General treatment group (Active Comparator): hot pack application on shoulder region upper trapezius massage two stretching exercises (modified sleeper stretch and modified cross-body stretch)
  Interventions: Other: Stretching exercises; Other: Hot pack; Other: Massage

INTERVENTIONS:
Other: Eccentric-focused exercises — Three eccentric-focused exercises:
  1. Shoulder external rotator eccentric contraction in shoulder abduction 90 degree
  2. Shoulder external rotator eccentric contraction in shoulder abduction 0 degree
  3. Shoulder abductor eccentric contraction in shoulder abduction 90 degree
  Arms: Eccentric-focused exercise group
Other: Stretching exercises — 1. Modified sleeper stretch
  2. Modified cross-body stretch
Other: Hot pack — Hot pack application on shoulder region
Other: Massage — Massage for upper trapezius

SUMMARY:
The aim of this study is to investigate the effects of shoulder eccentric exercise training on shoulder mobility, rotator cuff strength, pain and dysfunction, scapular kinematics and muscle activation in symptomatic overhead athletes with posterior shoulder tightness.

DETAILED DESCRIPTION:
Overhead athletes commonly have posterior shoulder tightness due to repetitively high tensile loading during overhead throwing. However, intervention studies focused on posterior shoulder tightness in people with subacromial pain are still limited. Additionally, eccentric exercise was thought to improve the eccentric strength and neuromuscular control of posterior shoulder muscles to endure repetitively eccentric loading, which may improve posterior shoulder tightness and decrease the risk of subacromial pain. Nevertheless, no previous study investigated the influence of eccentric exercise on posterior shoulder tightness in overhead athletes. The aim of this study is to investigate the effects of shoulder eccentric exercise training on shoulder mobility, rotator cuff strength, pain and dysfunction, scapular kinematics and muscle activation in symptomatic overhead athletes with posterior shoulder tightness.

ELIGIBILITY:
Inclusion Criteria:

* Participate in overhead sports over 4 hours per week
* Age between 20 to 50 years old
* Glenohumeral joint range of motion deficit: Shoulder internal rotation loss more than 15 degrees compared to the non-dominant side and total arc of motion loss more than 5 degrees or/and horizontal adduction range of motion lo more than 15 degrees compared to the non-dominant side
* Shoulder impingement syndrome criteria

Exclusion Criteria:

* History of shoulder dislocation, fracture and operation
* History of direct contact in upper extremities or cervical region in the past one month
* Shoulder pain or neurological symptom caused by cervical problem
* VAS more than 5 during shoulder elevation
* Receive treatment for posterior shoulder tightness in the past 3 months

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11-09 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Shoulder range of motion (measured with goniometer) | 4 weeks
  Shoulder external rotation, internal rotation, horizontal adduction range of motion in shoulder flexion 90 degrees
Rotator cuff functional strength ratio (Pro 4, Biodex Medical Systems, Inc., Shirley, NY, USA) | 4 weeks
  Eccentric strength of shoulder external rotator and concentric strength of shoulder internal rotator are measured with isokinetic
Shoulder pain | 4 weeks
  Pain is measured with Visual Analogue scale (VAS) Score range from 0 to 10. Scoring of 0 represents no pain and scoring of 10 represents pain as bad as it could possibly be.
Shoulder function | 4 weeks
  Shoulder function is measured with Disability of the Arm, Shoulder and Hand questionnaire (DASH) Score range from 0 to 100. The higher of the score, the more disability.
Shoulder endurance test | 4 weeks
  Participants will be instructed to execute a shoulder endurance test with the theraband®. Participants are asked to place their tested arm in a shoulder forward flexion 90-degree position, holding a 1-m long theraband® fixed at shoulder height on a graduated stick. Then, they are asked to pull the theraband® from the starting position to a 90-90 ending position at an alternated cadence given by a metronome. Males were asked to pull a green theraband® (2.1 kg) and females a red theraband ® (1.7 kg).

SECONDARY OUTCOMES:
Electromagnetic tracking system (Liberty electromagnetic tracking system, Polhemus , Colchester, VT,) | 4 weeks
  Scapular kinematics during shoulder elevation task in scapular plane
Surface electromyography (TeleMyo 2400T G2, Noraxon USA Inc., Scottsdale, AZ, USA) | 4 weeks
  Muscle activation of infraspinatus, upper trapezius, lower trapezius and serratus anterior during shoulder elevation task in scapular plane

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Beitou, Taiwan